CLINICAL TRIAL: NCT07149155
Title: Adapting Stress First Aid (SFA) to the Needs of Harm Reduction Workers (HRWs) Serving Persons Who Use Drugs (PWUD) - Training and Pilot Testing Phase (Aim 2 and Aim 3)
Brief Title: Adaptation of SFA for HRW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00006228; R61DA059887 (NIH)
Record Dates: First submitted 2025-08-18; First posted 2025-08-29 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-08

CONDITIONS: Occupational Health
Keywords: Stress First Aid; Harm Reduction Workers; Persons who use drugs; overdose prevention; community outreach workers; peer workers

STUDY DESIGN:
Intervention Model Description: Pilot test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stress First Aid (Experimental): Harm Reduction Workers received Stress First Aid training and learning collaboratives
  Interventions: Behavioral: Stress First Aid for Harm Reduction Workers

INTERVENTIONS:
Behavioral: Stress First Aid for Harm Reduction Workers — The intervention was a 2-hour, in-person SFA/HRW training followed by 30-minute monthly learning collaboratives to address occupational stress of harm reduction workers.
  Other Names: SFA/HRW

SUMMARY:
The aim of this study is to pilot and test the feasibility, acceptability, and effectiveness of a Stress First Aid (SFA) intervention adapted for Harm Reduction Workers (HRWs) serving Persons Who Use Drugs. The intervention consists of a training and learning collaboratives used to reinforce the SFA principles

ELIGIBILITY:
Inclusion Criteria:

* Legal age of majority (18 +),
* Ability to read and speak conversational English, and
* Work as an HRW in substance misuse.

Exclusion Criteria:

* Inability to provide consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-09-24 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 24 2024 - October 1 2024 in harm reduction organization
Groups:
- Stress First Aid: Harm Reduction Workers received 2-hour in-person Stress First Aid (SFA) training and four, 30-minute learning collaboratives to reinforce SFA core components.
Period: Overall Study
Arm/Group | Stress First Aid
Started | 35
Completed | 25
Not Completed | 10
Not completed — Lost to Follow-up | 10

BASELINE CHARACTERISTICS:
Arm/Group | Stress First Aid
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.52 (10.93)
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 22
  More than one race | 3
  Unknown or Not Reported | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 3
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 22
  Male | 10
  Unknown or Not Reported | 3
Baseline Mean Knowledge of Stress First Aid (SFA) [Mean (Standard Deviation); unit: Score on a Scale] — A 3-item, 5-point Likert type sub-scale of Stress First Knowledge, Confidence, and Beliefs Scale, developed by the developers of Stress First Aid (SFA), with a minimum score 1 "Does not describe me at all", maximum score 5 "Describes me very well", where a higher score is a better outcome. Population: Two participants did not complete a baseline assessment.
  Score on a Scale
    number analyzed (Participants) | 33
    (all) | 3.15 (0.61)
Baseline Mean Confidence in Stress First Aid (SFA) [Mean (Standard Deviation); unit: Score on a Scale] — A 6-item, 5-point Likert type sub-scale of Stress First Knowledge, Confidence, and Beliefs Scale, developed by the developers of Stress First Aid (SFA), with a minimum score 1 "Does not describe me at all", maximum score 5 "Describes me very well", where a higher score is a better outcome. Population: Two participants did not complete a baseline assessment.
  Score on a Scale
    number analyzed (Participants) | 33
    (all) | 3.06 (0.63)
Baseline Mean Beliefs in Stress First Aid (SFA) [Mean (Standard Deviation); unit: Score on a Scale] — A 5-item, 5-point Likert type sub-scale of Stress First Knowledge, Confidence, and Beliefs Scale, developed by the developers of Stress First Aid (SFA), with a minimum score 1 "Does not describe me at all", maximum score 5 "Describes me very well", where a higher score is a better outcome. Population: Two participants did not complete a baseline assessment.
  Score on a Scale
    number analyzed (Participants) | 33
    (all) | 3.93 (0.58)

OUTCOME MEASURES:

1. Primary Outcome: Mean Knowledge of Stress First Aid (SFA) Assessed by Stress First Aid Knowledge, Confidence, and Beliefs - Knowledge Sub-Scale at 4 Months
Description: A 3-item, 5-point Likert type sub-scale of Stress First Knowledge, Confidence, and Beliefs Scale, developed by the developers of Stress First Aid (SFA), with a minimum score 1 "Does not describe me at all", maximum score 5 "Describes me very well", where a higher score is a better outcome.
Time Frame: Assessed from enrollment to the end of the intervention at 4 months, 4 months reported
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Stress First Aid
Number analyzed (Participants) | 25
Score on a Scale | 4.01 (0.54)

2. Primary Outcome: Mean Confidence in Stress First Aid (SFA) Assessed by Stress First Aid Knowledge, Confidence, and Beliefs - Confidence Sub-Scale at 4 Months
Description: A 6-item, 5-point Likert type sub-scale of Stress First Knowledge, Confidence, and Beliefs Scale, developed by the developers of Stress First Aid (SFA), with a minimum score 1 "Does not describe me at all", maximum score 5 "Describes me very well", where a higher score is a better outcome.
Time Frame: Assessed from enrollment to the end of the intervention at 4 months, 4 months reported
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Stress First Aid
Number analyzed (Participants) | 25
Score on a Scale | 3.90 (0.56)

3. Primary Outcome: Mean Beliefs in Stress First Aid (SFA) Assessed by Stress First Aid Knowledge, Confidence, and Beliefs - Beliefs Sub-Scale at 4 Months
Description: A 5-item, 5-point Likert type sub-scale of Stress First Knowledge, Confidence, and Beliefs Scale, developed by the developers of Stress First Aid (SFA), with a minimum score 1 "Does not describe me at all", maximum score 5 "Describes me very well", where a higher score is a better outcome.
Time Frame: Assessed from enrollment to the end of the intervention at 4 months, 4 months reported
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Stress First Aid
Number analyzed (Participants) | 25
Score on a Scale | 4.26 (0.41)

4. Primary Outcome: Mean Acceptability of SFA Assessed by Acceptability of Intervention Measure (AIM)
Description: A 4-item, 5-point Likert-type scale from Weiner et al., 2017, with a minimum score 1 "Completely disagree", maximum score 5 "Completely agree", where a higher score is a better outcome.
Time Frame: Immediately after the 2-hour, in-person training.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Stress First Aid
Number analyzed (Participants) | 30
Score on a Scale | 4.40 (0.79)

5. Primary Outcome: Mean Appropriateness of SFA Assessed by Intervention Appropriateness Measure (IAM)
Description: as for outcome 4
Time Frame: Immediately after the 2-hour, in-person training.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Stress First Aid
Number analyzed (Participants) | 30
Score on a Scale | 4.56 (0.80)

6. Primary Outcome: Mean Feasibility of SFA Assessed by Feasibility of Intervention Measure (FIM)
Description: as for outcome 4
Time Frame: Immediately after the 2-hour, in-person training.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Stress First Aid
Number analyzed (Participants) | 30
Score on a Scale | 4.45 (0.58)

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed and the reason the number who were at risk was zero is because this was a benign behavioral intervention that was educational in nature.
Arm/Group | Stress First Aid
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-09-13): https://cdn.clinicaltrials.gov/large-docs/55/NCT07149155/Prot_000.pdf
  • Informed Consent Form (2024-09-13): https://cdn.clinicaltrials.gov/large-docs/55/NCT07149155/ICF_001.pdf